CLINICAL TRIAL: NCT01177930
Title: Evaluation of the Health Related Quality of Life and Disease Prevalence of Children From Spain at 6-8 Years of Age Who Participated in a Qualifying Infant Formula Study at Birth
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Other Study IDs: 6004
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Feeding with milk with DHA and ARA
- Feeding with milk without DHA and ARA

SUMMARY:
The purpose of this study is to evaluate the influence of the type of feeding in the first year of life on the behavior and health-related quality of life at 6-8 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Father, mother or legal representative of a child who was included in the qualifying study
* Child 6 - 8 years of age
* Written informed consent of the father, mother or legal representative

Exclusion Criteria:

* None

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 6 - 8 years of age
Sampling Method: Non-Probability Sample
Dates: Start 2009-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Influence of the type of feeding from the first year of life on the quality of life in the same children at 6 - 8 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- E-C-Bio, S.L., Las Rozas de Madrid, Madrid, Spain